CLINICAL TRIAL: NCT04911010
Title: Effectiveness of Trauma Therapy Using Prolonged Exposure for the Treatment of Post-traumatic Stress Disorder (PTSD) in Patients With Comorbid Psychotic Disorder
Brief Title: Effectiveness of Trauma Therapy in Patients With PTSD and Comorbid Psychotic Disorder
Acronym: PEPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Susanne Sarkar, Dr. Susanne Sarkar, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHH-HSA-PEPSY
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Post Traumatic Stress Disorder; Psychotic Disorders; Psychosis; Schizophrenia; PTSD
Keywords: PEPSY; Prolonged Exposure; trauma psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, parallel-group, two-armed, multicentre, open trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Prolonged Exposure + Treatment as usual (Experimental): Participants in this arm will receive 16 weekly sessions with Prolonged Exposure Therapy (RT) over 4 months in addition to their treatment as usual.
  Interventions:
  Behavioral: Prolonged Exposure Therapy Other: Treatment as usual
  Interventions: Behavioral: Prolonged Exposure
- Waiting-Controll-Group (No Intervention): Treatment as usual Treatment as usual will include medication management, supportive brief counselling sessions and various types of psychosocial (e.g. social work guided support, peer support) and monitoring provided by Mental Health Services, with individual and family psychological therapies offered occasionally.
  Intervention: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Prolonged Exposure — In the intervention condition, patients are treated with prolonged exposure in 16 hours of individual therapy immediately after the baseline measurement. The 16 individual therapeutic sessions take place 1 to 2 sessions per week over a period of 7 to 16 weeks. The individual therapeutic sessions are recorded on video with camera focus on the therapist. Parts of the prolonged exposure procedure (reliving the traumatic memory) are recorded on tape (via the patient's personal smartphone) so that the patient can listen to the recording as homework at home. The patients then take part in a post-treatment study diagnosis (T1).
  Other Names: Trauma Therapy
  Arms: Experimental: Prolonged Exposure + Treatment as usual

SUMMARY:
Effectiveness of trauma therapy using prolonged exposure for the treatment of post-traumatic stress disorder (PTSD) in patients with comorbid psychotic disorder

DETAILED DESCRIPTION:
Background and goals: Patients with psychotic disorders often report traumatizing experiences in their biography and show symptoms of a trauma-related disorder. It is assumed that around 30 percent of patients with a psychotic disorder also meet the criteria for PTSD. For the vast majority of patients, psychosis is the focus of mostly pharmacological treatment, while PTSD is not part of the therapy. In a first randomized controlled study, van den Berg's Dutch working group was able to show that psychosis patients with comorbid PTSD who were given a classic trauma exposure procedure showed a high response to PTSD symptoms (van den Berg et al., 2015). It is also important that in this study the trauma exposure did not lead to an increase in psychotic symptoms or undesirable side effects (e.g. suicidality). In order to examine the question of the generalizability of the effects, a randomized controlled study in the German-speaking health care system is necessary. In the following efficacy study in which psychosis patients with PTSD are treated using prolonged exposure. METHODS AND RESULTS: It is a multicenter, controlled, prospective, randomized study (RCT). It is investigated whether trauma therapy reduces PTSD and psychosis symptoms compared to the Treatment-As-Usual Waiting Group (TAU). The primary endpoint is the severity of the PTSD symptoms between the baseline measurement and the 6-month follow-up. Secondary endpoints are subjective PTSD symptoms, paranoia, hallucinations, and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of a Post Traumatic Stress Disorder (PTSD spectrum disorder (ICD-10, F43.1, confirmed by SCID-5 and CAPS)
* have a diagnosis of a schizophrenia spectrum disorder (ICD-10, F2, confirmed by SCID-5)
* patients will be reporting distressing AH for at least six months (to be beyond the startle and adjustment phase ) and score ≥ 3 on either item 8 or item 9 of the PSYRATS-AH;
* be ≥ 18 years of age
* good knowledge of the German language
* Willingness to participate in randomization and trauma-focused therapy

Exclusion Criteria:

* Changes in neuroleptic or antidepressant therapy within the last 4 weeks (exclusion of drug effects)
* Any substance addiction with continued use other than nicotine and / or caffeine addiction
* IQ of 70 or less
* Acute suicidality
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS) | 6 months after baseline assessment
  The severity of the PTSD symptoms associated distress. The distress factor score of the CAPS is the primary outcome as this is what has been prioritized by patients and is relevant to functioning. Confirmatory analysis will be conducted based on the intent-to-treat population (ITT), defined on the basis of the ITT principle. The aim is to show that the intervention group is superior to the control meaning that the mean score at 6 months adjusted for the baseline value is lower in the intervention group than in the control group. Lower scores indicate less distress.
Subjective PTSD symptoms | 6 months after baseline assessment
  Posttraumtatic Stress Symptom Scale Self-Report (PSSI, Foa et al., 1993)

SECONDARY OUTCOMES:
The Psychotic Symptom Rating Scales-AH-Distress factor score (PSYRATS-AH) | 6 months after baseline assessment
  Auditory hallucination associated distress. The distress factor score of the PSYRATS-AH is the secondary outcome. The aim is to show that the intervention group is superior to the control meaning that the mean score at 6 months adjusted for the baseline value is lower in the intervention group than in the control group. Lower scores indicate less distress.
Welleing | 6 months after baseline assessment
  Wellbeing: Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, NHS Health Scotland, University of Warwick and University of Edinburgh, 2007)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided